CLINICAL TRIAL: NCT01073878
Title: Athena PMT - Device to Treat Urinary Incontinence - Effectiveness, Tolerability and Satisfaction "Athena D.U.E.T.S. Trial"
Brief Title: Athena Pelvic Muscle Trainer - DUETS Trial
Acronym: DUETS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Athena Feminine Technologies, Inc. (Industry)
Responsible Party: David M. Berryman, Athena FT
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PMT-4-001
Record Dates: First submitted 2010-02-17; First posted 2010-02-23 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Urinary Incontinence
Keywords: Urinary Urge Incontinence; Urinary Stress Incontinence; Urinary Mixed Incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Athena Pelvic Muscle Trainer — The Athena PMT is a vaginally inserted electrical stimulator that induces the pelvic floor muscles to contract and relax, similar to Kegel exercises intended to strengthen the pelvic floor muscles.
  Other Names: Athena PMT; PMT; Pelvic Muscle Trainer; Athena

SUMMARY:
The purpose of this study is to determine if the Athena Pelvic Muscle Trainer device effectively treats stress, urge or mixed incontinence in women by strengthening the pelvic floor muscles by collecting data from the patient on the

1. Over Active Bladder Questionnaire
2. The 7-Day Urine Diary questionnaire

   This study will also look at whether or not there is an improvement in sexual health after using the device by collecting data frm the patient on the
3. Female Sexual Function Index questionnaire

DETAILED DESCRIPTION:
This is a Phase IV, prospective, open-label, multi-center, observational study to assess the effectiveness of the Athena PMT to relieve or eliminate the symptoms of female urinary incontinence.

The study will enlist approximately 100 or more Nurse-Practitioners in Women's Health as the principle investigators from community-based primary care centers (OB-GYN, Internal Medicine, Family Practices or Women's Health Centers) who will enroll approximately 500 or more subjects who suffer from urge and/or stress urinary incontinence and who may benefit from strengthening of Kegel muscles of the pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 30 and 70 years
2. Suffer from urge-incontinence, stress incontinence or incontinence of mixed etiology and who may benefit from strengthening Kegel muscles by electrical stimulation
3. Able to provide informed consent and physically able to comply with protocol requirements.
4. Experience one or more incontinence episodes per week.
5. Women of childbearing potential must have a negative urine or blood pregnancy test within 7 days prior to initiation of treatment.
6. Subject may be post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (e.g., hormonal contraceptive, intra- uterine device (IUD), diaphragm with spermicide, condom with spermicide or abstinence) from the screening visit through the duration of study participation.
7. Have a positive response to two or more questions on the Athena Questionnaire

Exclusion Criteria:

1. Neurological deficiency that does not permit proper sensory perception or stimulation.
2. Is currently pregnant, lactating or attempting to get pregnant
3. Has a cardiac pacemaker or a history of rate or conductive disturbance
4. Has anatomical vaginal structures that do not permit proper and complete placement of the trainer.
5. Has irregular menstrual bleeding cycles.
6. Has urinary or vaginal infections, localized lesions, or other undiagnosed symptoms.
7. Has a history or symptoms of urinary retention.
8. Has cancer or a life expectancy of less than one year
9. Recreational drug use
10. Consume more than three caffeine beverages daily
11. Consume more than 1-2 alcoholic drinks per day
12. Significant drug use (causing diuresis or urinary retention
13. Allergy or sensitivity to materials in the Athena PMT
14. Participation in another clinical trial within past 3 months
15. Subjects morbidly obese (BMI >35)
16. Subjects who chronically smoke (> 10 cigarettes per day)
17. Subjects required to do heavy lifting (> 40 pounds regularly)
18. Surgery within the past six months for incontinence, or use of other incontinence devices
19. Currently taking cholinergic or anti-cholinergic drugs or other prescription or non-prescription drugs that may increase or decrease the volume or frequency of urination and thus, may confound the results of this study, except, in the opinion of the investigator. The subject's regimen has been stable for at least sixty days.
20. Suspected infection or condition (e.g., diabetes) that would alter the subjects ability to participate or would confound the results of the trial

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To assess objective treatment outcomes of urge, stress or mixed incontinence. | 5 Visits over 13 weeks. Subjects are seen in the office at Screening Visit 1 (Week -1), Visit 1a (Week 0), Visit 2 (Week 2), Visit 3 (Week 6), Visit 4 (Week 12)
  Outcomes will be measured via patient questionnaires over a 13 week trial. Visit 1 (Week -1) and Visit 4 (Week 12) values for the Overactive Bladder Questionnaire and the Female Sexual Function Index will be captured. 7-day Urine Diaries will be captured for the week preceeding visits 2, 3 and 4.

SECONDARY OUTCOMES:
Evaluate effectiveness, tolerability, satisfaction and compliance of the Athena PMT across a wide demographic population using: 1) the Subject Satisfaction Evaluation questionnaire | At Visit 4 (Week 12)
  At the last visit, patients will complete a Subject Satisfaction Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Shaw, MD, Study Director — Director of Women's Health, Yale University
Locations (97):
- United States (96):
  - John Foster MD, Birmingham, Alabama
  - La Mamma Spa, Birmingham, Alabama
  - Kyle Chavers MD, Dothan, Alabama
  - Salud! for Women, Casa Grande, Arizona
  - New Horizons Women's Care, Chandler, Arizona
  - Barbara Wiggin PhD, ANP-C, Peoria, Arizona
  - Agnes Oblas APRN, Phoenix, Arizona
  - Arcadia Well Woman, Scottsdale, Arizona
  - Patricia A Faust, Tempe, Arizona
  - Beth Andresen, Tucson, Arizona
  - Teresa Mote RNC NP, Tucson, Arizona
  - Brenda Hanson-Smith, RN, DNS, OGNP, El Dorado Hills, California
  - Lynda Reed, Ontario, California
  - Rose Mary Mosher, Rolling Hills Est., California
  - Evan Vapnek MD, San Diego, California
  - Marilyn Brooks, San Jacinto, California
  - Healthworks, San Luis Obispo, California
  - Maureen Allen, Northglenn, Colorado
  - Kristan Langdon, ANP-C, Parker, Colorado
  - Karen D. Adamson, Salida, Colorado
  - Merrilyn H. McNatt APRN, New London, Connecticut
  - Jean Ohliger APRN, South Windsor, Connecticut
  - Arlena Falcon, Blountstown, Florida
  - Carl Spirazza, Boynton Beach, Florida
  - Khadra Mohamoud Osman mD, Fort Lauderdale, Florida
  - Shelly E Kramer ARNP, Lake Worth, Florida
  - Ivonne M. Reynolds, Margate, Florida
  - Susan Chappuis, ARNP-C, Ormond Beach, Florida
  - Elizabeth Tsarnas, Stuart, Florida
  - Bayside Gynecology, P.A., Venice, Florida
  - Jeffrey C Seiler, MD, West Palm Beach, Florida
  - Deborah Cothran WHNP-BC, Albany, Georgia
  - Elizabeth Killebrew MD, Fayetteville, Georgia
  - Michael D Benson, Deerfield, Illinois
  - Laurie Knoke, DeKalb, Illinois
  - Sherry Owen, APN, Gurnee, Illinois
  - Julie Snow, Park Ridge, Illinois
  - Kathryn A. Copeland, Carmel, Indiana
  - Matthew Sprunger MD, Fort Wayne, Indiana
  - Tamara Meisel ARNP, Lakin, Kansas
  - Richard F. Ford MD, Ashland, Kentucky
  - Women's Care Center, Lexington, Kentucky
  - Tammi K Herkey, Bossier City, Louisiana
  - Stefanie A Schultis, Covington, Louisiana
  - Steven Lenowitz, MD, Bel Air, Maryland
  - Kathryn Cervi, Columbia, Maryland
  - Elizabeth P Sipala, Galena, Maryland
  - Deborah A. Davis, MSN, CRNP, Prince Frederick, Maryland
  - Martha Klay, Great Barrington, Massachusetts
  - Pioneer Valley Urology, Springfield, Massachusetts
  - Margaret Duggan, Walpole, Massachusetts
  - Kathryn Koches, Dearborn, Michigan
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Isabel M Raposo, Riverview, Michigan
  - Laura Hintz, Saginaw, Michigan
  - Mickie G. Autry PhD, NP-C, Jackson, Mississippi
  - Kathleen M. Young RNC NP, Kalispell, Montana
  - Urogynecology Arts of New Jersey, East Brunswick, New Jersey
  - Lynda M. Adamson, Galloway, New Jersey
  - Women's Total Health, Hamburg, New Jersey
  - Cindy Nevara APN, Vineland, New Jersey
  - Jeanne Ann Dahl, RNC, WHNP, Albany, New York
  - Meredith Schledorn, Cortland, New York
  - Raj Mahajan MD, Oswego, New York
  - Diane Stonemetz, West Seneca, New York
  - Kathy Edwards, Minot, North Dakota
  - Columbus OB/Gyn Inc., Columbus, Ohio
  - Holly Murphy, Columbus, Ohio
  - Susan Frost, Columbus, Ohio
  - Amy G Brenner M.D, Fairfield, Ohio
  - Elizabeth D. Allen CNP, Gallipolis, Ohio
  - William Shuler, MD, Tulsa, Oklahoma
  - Deborah Malone, Bend, Oregon
  - Anne Marie Moore, Womens Health Nurse Practitioner, Eugene, Oregon
  - Cathleen Ann Folk FNP, Portland, Oregon
  - Mary L Hagood, FNP-C, Roseburg, Oregon
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania
  - Paulette Schreiber, CRNP, Saint Mary's, Pennsylvania
  - Marie T Ziegler, West Chester, Pennsylvania
  - Nancy Newman RNC, WHNP, Lexington, South Carolina
  - Sharon Little, Collierville, Tennessee
  - Margaret A. Hull, Franklin, Tennessee
  - Urology Associates, P.C., Nashville, Tennessee
  - John Pickel MD, Arlington, Texas
  - Christopher J. Jayne, MD, FACOG, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Marney Kidwell RNC, San Antonio, Texas
  - D. Crawford Allison MD, Waco, Texas
  - Laura C. Maw, Lehi, Utah
  - Betsy Browning, Bennington, Vermont
  - Anne L Stephens, Chesapeake, Virginia
  - Rand Gynecology, LLC, Chesapeake, Virginia
  - Julie Spencer, Lansdowne, Virginia
  - Patrice C Malena, Newport News, Virginia
  - Ocean Beach Women's Clinic, Ilwaco, Washington
  - Kimberly Scheer, Vashon, Washington
- Primary Care, PLLC, Christiansted, VI, Virgin Islands